CLINICAL TRIAL: NCT04789993
Title: Additional Autoimmune Diseases With Type 1 Diabetes in Children and Adolescents at Diabetes Diagnostic and During Follow-up : a Monocentric Study in France
Brief Title: Additional Autoimmune Diseases With Type 1 Diabetes in Pediatrics at Diabetes Diagnosis and During Follow-up
Acronym: AADT1D
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LEGAGNEUR Carole, MD, Central Hospital, Nancy, France
Other Study IDs: 2020PI283
Record Dates: First submitted 2021-02-20; First posted 2021-03-10 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Type 1 Diabetes; Autoimmune Diseases; Hashimoto Disease; Graves Disease; Celiac Disease; Addison Disease; Vitiligo
Keywords: Type 1 diabetes; Autoimmune Diseases; Pediatrics; Children; Adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases; Hashimoto Disease; Graves Disease; Celiac Disease; Addison Disease; Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. — There is no intervention needed. It is a retrospective cohort. The usual follow-up of type 1 diabetes is studied from its beginning to the last news of the patient.

SUMMARY:
This study aims to describe the prevalence of additional autoimmune diseases and their specific antibodies at type 1 diabetes (T1D) diagnosis, and their incidence rate during follow-up, for children and adolescents. It also aims to describe the characteristics of the pediatric cohort followed since 2014 for type 1 diabetes by one of France's centers of reference for paediatric diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes diagnosed with the following criteria: (i) Classic symptoms of diabetes or hyperglycemic crisis, with plasma glucose concentration ≥11.1 mmol/L (200 mg/dl), or (ii) fasting plasma glucose ≥7.0 mmol/l (≥126 mg/dl) ; and (iii) presence of diabetes associated autoantibodies : ICA, GAD, IA2, IAA and/or ZnT8
* age < 18 years old at type 1 diabetes diagnostic
* type 1 diabetes diagnosed between 2014-01-01 and 2021-02-01

Exclusion Criteria:

* type 1 diabetes diagnostic not certain

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patient followed for type 1 diabetes at the Children's Hospital of Nancy, France, between 2014-01-01 and 2021-02-01.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of additional autoimmune diseases at type 1 diabetes diagnosis | up to 3 weeks after type 1 diabetes diagnosis
  Will be studied the additional autoimmune diseases to type 1 diabetes listed in the 2018 ISPAD recommendations
Type of additional autoimmune diseases at type 1 diabetes diagnosis | up to 3 weeks after type 1 diabetes diagnosis
  Will be studied the additional autoimmune diseases to type 1 diabetes listed in the 2018 ISPAD recommendations

SECONDARY OUTCOMES:
Characteristics of patients, if additional autoimmune disease is present or absent | up to 3 weeks after type 1 diabetes diagnosis
  Family and personal history, biological, serological, anthropometrical characteristics at type 1 diabetes diagnostic
Occurence or non-occurence of at least one additional autoimmune diseases during follow-up | From type 1 diabetes diagnostic to last news date, an average of 3 years
  Will be studied the additional autoimmune diseases to type 1 diabetes listed in the 2018 ISPAD recommendations
Occurence or non-occurence of each type of additional autoimmune disease during follow-up | From type 1 diabetes diagnostic to last news date, an average of 3 years
  Will be studied the additional autoimmune diseases to type 1 diabetes listed in the 2018 ISPAD recommendations, in this outcome studied each one separately
Presence of antibodies specific to an additional autoimmune disease at type 1 diabetes diagnostic | up to 3 weeks after type 1 diabetes diagnosis
  Antibodies detected in the serum, antibodies specific to the following autoimmune diseases : Hashimoto (Thyroid peroxidase antibodies, and/or thyroglobulin antibodies) Graves disease (TRAK), coeliac disease (anti-tissue transglutaminase (tTG) antibodies,endomysial antibodies (EMA)), Addison disease ( adrenal antibodies ), autoimmune gastritis (parietal cell antibodies)
Characteristics of patients, if at least one type of antibodies specific to an autoimmune disease is present or absent at type 1 diabetes diagnostic | up to 3 weeks after type 1 diabetes diagnosis
  Family and personal history, biological, serological, anthropometrical characteristics at type 1 diabetes diagnostic
Characteristics of patients, for each type of antibodies specific to an autoimmune disease, present or absent at type 1 diabetes diagnostic | up to 3 weeks after type 1 diabetes diagnosis
  Family and personal history, biological, serological, anthropometrical characteristics at type 1 diabetes diagnostic
Occurence or non-occurence of at least one type of antibody specific to an additional autoimmune disease | From type 1 diabetes diagnosis to last news date, from 1 to 6 years
  Antibodies detected in the serum, antibodies specific to the following autoimmune diseases : Hashimoto (Thyroid peroxidase antibodies, and/or thyroglobulin antibodies) Graves disease (TRAK), coeliac disease (anti-tissue transglutaminase (tTG) antibodies,endomysial antibodies (EMA)), Addison disease ( adrenal antibodies ), autoimmune gastritis (parietal cell antibodies)
Occurence or non-occurence of antibodies specific to each additional autoimmune disease listed in outcome 5 | From type 1 diabetes diagnosis to last news date, from 1 to 6 years
  Antibodies detected in the serum, antibodies specific to the following autoimmune diseases : Hashimoto (Thyroid peroxidase antibodies, and/or thyroglobulin antibodies) Graves disease (TRAK), coeliac disease (anti-tissue transglutaminase (tTG) antibodies,endomysial antibodies (EMA)), Addison disease ( adrenal antibodies ), autoimmune gastritis (parietal cell antibodies)
Description of the characteristics of all the patients followed in our cohort of pediatric type 1 diabetes | Up to 3 weeks after type 1 diabetes diagnosis
  Family and personal history, biological, serological, anthropometrical characteristics at type 1 diabetes diagnostic, presence of antibodies specific to an additional autoimmune disease, and occurence of additional autoimmune diseases
Description of the autoimmune characteristics of all the patients followed in our cohort of pediatric type 1 diabetes | during follow-up : From type 1 diabetes diagnosis to last news date, from 1 to 6 years
  presence of antibodies specific to an additional autoimmune disease, and occurence of additional autoimmune diseases
If detection of antibodies specific to an additional autoimmune disease : delay between detection of these antibodies and diagnosis of the corresponding autoimmune disease | From type 1 diabetes diagnosis to last news date, from 1 to 6 years
  Antibodies detected in the serum, antibodies specific to the following autoimmune diseases : Hashimoto (Thyroid peroxidase antibodies, and/or thyroglobulin antibodies) Graves disease (TRAK), coeliac disease (anti-tissue transglutaminase (tTG) antibodies,endomysial antibodies (EMA)), Addison disease ( adrenal antibodies ), autoimmune gastritis (parietal cell antibodies)
If patient diagnosed with Hashimoto when type 1 diabetes is diagnosed, proportion of patients with thyroid dysfunction | Up to 3 weeks after type 1 diabetes diagnosis
  Thyroid dysfunction : hormonal dysfunction associated to Hashimoto
Occurence of thyroid dysfunction in patients with type 1 diabetes and Hashimoto | From type 1 diabetes diagnosis to last news date, from 1 to 6 years
  Occurence during type 1 diabetes follow-up of thyroid dysfunction in patients with Hashimoto
Proportion of patients with thyroid dysfunction due to Hashimoto needing a specific treatment | Up to 3 weeks after type 1 diabetes diagnosis
Occurence of specific treatment onset in patients followed for type 1 diabetes with thyroid dysfunction due to Hashimoto | From type 1 diabetes diagnosis to last news date, from 1 to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Carole LEGAGNEUR, MD, Study Director — Centre Hospitalo-Universitaire de Nancy, Hôpital d'Enfants de Brabois
Locations (1):
- Hôpital d'Enfants de Brabois, Vandœuvre-lès-Nancy, Lorraine, France